CLINICAL TRIAL: NCT00372424
Title: An Explorative Study Of The Tolerability Of SU011248 In Combination With Docetaxel And Trastuzumab As First-Line Treatment In Patients With Breast Cancer Over-Expressing HER-2
Brief Title: Study Of SU011248 In Combination With Docetaxel And Trastuzumab In Patients With Advanced Breast Cancer HER-2 Positive
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6181113
Record Dates: First submitted 2006-09-05; First posted 2006-09-07 (Estimated); Results first posted 2012-10-30 (Estimated); Last update posted 2012-12-28 (Estimated); Status verified 2012-12

CONDITIONS: Breast Cancer
Keywords: Breast cancer over-expressing HER2. First-line treatment with sunitinib/docetaxel/trastuzumab.
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Sunitinib; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Combination of SU011248 (37.5 mg once daily [Schedule 2/1]) with docetaxel (75 mg/m2 every 3 weeks) and trastuzumab (therapeutic dose)
  Interventions: Drug: Herceptin; Drug: Sunitinib; Drug: Taxotere

INTERVENTIONS:
Drug: Herceptin — Trastuzumab will be administered intravenously on Day 1 before docetaxel - loading dose of 4 mg/kg over 90-minute on Day 1 followed by weekly maintenance doses of 2 mg/kg on Days 1, 8, 15 given as 30-minute infusions if the initial loading dose was well tolerated. Loading dose of 8 mg/kg over 90-minute on Day 1 followed by 3-weekly maintenance doses of 6 mg/kg given as 90-minute infusions. The administration of 6 mg/kg will be repeated on Day 1 every 3 weeks.
  Other Names: trastuzumab
Drug: Sunitinib — SU011248 will be administered at 37.5 mg once daily for 2 weeks every 3 weeks (Schedule 2/1) starting from Day 2, when in combination with docetaxel. SU011248 will be administered at the starting dose of 37.5 mg daily in a continuous regimen when docetaxel is discontinued.
  Other Names: Sutent
Drug: Taxotere — The starting dose of docetaxel will be 75 mg/m2 every 3 weeks, administered on Day 1 of each cycle as a 1-hour IV infusion.
  Other Names: docetaxel

SUMMARY:
This is an exploratory trial evaluating the tolerability and preliminary anti-tumor activity of SU011248 combined with docetaxel and trastuzumab in patients with locally recurrent or metastatic breast cancer over-expressing Her-2, who have not received chemotherapy treatment in the advanced disease setting.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer with evidence of unresectable, locally recurrent, or metastatic disease.
* Tumors over-expressing Her-2
* Candidate for treatment with docetaxel/trastuzumab

Exclusion Criteria:

* Histology of inflammatory carcinoma
* AST and/or ALT >1.5 x ULN concomitant with ALP >2.5 x ULN

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2006-12; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- Belgium (4):
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Charleroi
  - Pfizer Investigational Site, Sint-Niklaas
  - Pfizer Investigational Site, Wilrijk
- Italy (2):
  - Pfizer Investigational Site, Meldola, FC
  - Pfizer Investigational Site, Milan

REFERENCES:
- [Derived] Cardoso F, Canon JL, Amadori D, Aldrighetti D, Machiels JP, Bouko Y, Verkh L, Usari T, Kern KA, Giorgetti C, Dirix L. An exploratory study of sunitinib in combination with docetaxel and trastuzumab as first-line therapy for HER2-positive metastatic breast cancer. Breast. 2012 Dec;21(6):716-23. doi: 10.1016/j.breast.2012.09.002. Epub 2012 Sep 27. PMID 23022045
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181113&StudyName=Study%20Of%20SU011248%20In%20Combination%20With%20Docetaxel%20And%20Trastuzumab%20In%20Patients%20With%20Advanced%20Breast%20Cancer%20HER-2%20Positive

RESULTS

PARTICIPANT FLOW:
Groups:
- Sunitinib + Docetaxel + Trastuzumab: Sunitinib 37.5 milligram (mg) capsule orally once daily continuously starting from Day 2 up to Day 15 in each cycle, in schedule 2/1 (2 week on treatment, 1 week off treatment) along with docetaxel 75 milligram/square meter (mg/m^2) intravenous infusion over 1 hour on Day 1 of each cycle and trastuzumab either weekly: loading dose of 4 milligram/kilogram (mg/kg) intravenous infusion over 90 minutes on Day 1 followed by weekly maintenance doses of 2 mg/kg intravenous infusion over 30 minutes; or every 3 weeks: loading dose of 8 mg/kg intravenous infusion over 90 minutes on Day 1 followed by maintenance doses of 6 mg/kg intravenous infusion over 90 minutes every 3 weeks. Cycle length was 3 weeks.
Period: Overall Study
Arm/Group | Sunitinib + Docetaxel + Trastuzumab
Started | 26
Treated | 25
Completed | 0
Not Completed | 26
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 1
Not completed — Death | 1
Not completed — Objective Progression or Relapse | 14
Not completed — Other | 7
Not completed — Enrolled, Not Treated | 1

BASELINE CHARACTERISTICS:
Arm/Group | Sunitinib + Docetaxel + Trastuzumab
Number analyzed (Participants) | 25
Age Continuous [Mean (Standard Deviation); unit: years] | 57.0 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A SAE was an AE resulting in any of following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: From screening until 28 days post last dose of study drug
Population: Safety population included all participants enrolled in the study who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Sunitinib + Docetaxel + Trastuzumab
Number analyzed (Participants) | 25
participants
  AEs | 24
  SAEs | 11

2. Secondary Outcome: Percentage of Participants With Objective Response (OR)
Description: Percentage of participants with objective response based assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). Confirmed responses are those that persist on repeat imaging study at least 4 weeks after initial documentation of response. CR are defined as disappearance of all target lesions. PR are those with at least 30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions.
Time Frame: Baseline, assessed every 6 weeks starting from Day1 of Cycle 3 up to end of treatment (Day 1344)
Population: Per protocol (PP) population included all participants who received at least 1 dose of sunitinib and had at least a tumor assessment post baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sunitinib + Docetaxel + Trastuzumab
Number analyzed (Participants) | 22
percentage of participants | 72.7 [49.8 to 89.3]

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Time in weeks from start of study treatment to first documentation of objective tumor progression or death due to any cause. PFS was calculated as (first event date minus the date of first dose of study medication plus 1) divided by 7. Tumor progression was determined from oncologic assessment data (where data meet the criteria for progressive disease [PD]), or from adverse event (AE) data (where the outcome was "Death").
Time Frame: Baseline, assessed every 6 weeks starting from Day1 of Cycle 3 up to end of treatment (Day 1344)
Population: Study population included all participants who received at least 1 dose of study medication.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Sunitinib + Docetaxel + Trastuzumab
Number analyzed (Participants) | 25
weeks | 58.4 [37.0 to 66.1]

4. Secondary Outcome: Duration of Response (DR)
Description: Time in weeks from the first documentation of objective tumor response to objective tumor progression or death due to any cancer. Duration of tumor response was calculated as (the date of the first documentation of objective tumor progression or death due to cancer minus the date of the first CR or PR that was subsequently confirmed plus 1) divided by 7. DR was calculated for the subgroup of participants with a confirmed objective tumor response.
Time Frame: Baseline, assessed every 6 weeks starting from Day1 of Cycle 3 up to end of treatment (Day 1344)
Population: Study population, subgroup of participants with a confirmed objective tumor response (CR or PR).
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Sunitinib + Docetaxel + Trastuzumab
Number analyzed (Participants) | 16
weeks | 51.3 [32.0 to 60.1]

5. Secondary Outcome: Plasma Trough Concentrations (Ctrough) of SU011248 (Sunitinib), SU012662 (Sunitinib Metabolite) and Total Drug (SU011248+SU012662)
Description: Ctrough = the concentration prior to study medication administration. Ctrough was calculated for SU011248 (Sunitinib), SU012662 (Sunitinib metabolite) and total drug (SU011248+SU012662). Concentration values below the lower limit of quantification were taken as zero.
Time Frame: Pre-dose (0 hours [H]) on Day 1 and Day 15 of Cycle 2, 4, 6 and additionally Day 15 of Cycle 1
Population: Pharmacokinetic (PK) analysis set included participants from study population who had completed sampling for pharmacokinetic profiles for study medication. 'n' is number of participants who were evaluable at given time points.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Sunitinib + Docetaxel + Trastuzumab
Number analyzed (Participants) | 25
nanogram/milliliter (ng/mL)
  Sunitinib: Cycle1/Day15 (n= 19) | 40.17 (32.17)
  Sunitinib: Cycle2/Day1 (n= 17) | 5.96 (6.17)
  Sunitinib: Cycle2/Day15 (n= 16) | 37.29 (31.07)
  Sunitinib: Cycle4/Day1 (n= 17) | 5.26 (5.71)
  Sunitinib: Cycle4/Day15 (n= 16) | 43.21 (27.31)
  Sunitinib: Cycle6/Day1 (n= 16) | 3.36 (4.34)
  Sunitinib: Cycle6/Day15 (n= 13) | 28.46 (21.19)
  Sunitinib Metabolite: Cycle1/Day15 (n= 19) | 16.15 (12.09)
  Sunitinib Metabolite: Cycle2/Day1 (n= 17) | 4.76 (3.92)
  Sunitinib Metabolite: Cycle2/Day15 (n= 16) | 14.43 (11.34)
  Sunitinib Metabolite: Cycle4/Day1 (n= 17) | 3.95 (2.57)
  Sunitinib Metabolite: Cycle4/Day15 (n= 16) | 17.62 (11.17)
  Sunitinib Metabolite: Cycle6/Day1 (n= 16) | 2.96 (2.89)
  Sunitinib Metabolite: Cycle6/Day15 (n= 13) | 11.54 (9.66)
  Total Drug: Cycle1/Day15 (n= 19) | 56.31 (42.70)
  Total Drug: Cycle2/Day1 (n= 17) | 10.72 (9.80)
  Total Drug: Cycle2/Day15 (n= 16) | 51.72 (41.45)
  Total Drug: Cycle4/Day1 (n= 17) | 9.21 (7.97)
  Total Drug: Cycle4/Day15 (n= 16) | 60.83 (37.43)
  Total Drug: Cycle6/Day1 (n= 16) | 6.32 (7.02)
  Total Drug: Cycle6/Day15 (n= 13) | 40.00 (30.04)

6. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Docetaxel
Description: Concentration values below the lower limit of quantification were taken as zero.
Time Frame: End of infusion (1 H) on Day 1 of Cycle 1, 2, 4 and 6
Population: PK analysis set included participants from study population who had completed sampling for pharmacokinetic profiles for study medication. 'n' is number of participants who were evaluable at given time points.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sunitinib + Docetaxel + Trastuzumab
Number analyzed (Participants) | 25
ng/mL
  Cycle1/Day1 (n= 23) | 1117.05 (1159.53)
  Cycle2/Day1 (n= 19) | 1388.63 (1260.94)
  Cycle4/Day1 (n= 16) | 1316.88 (1096.97)
  Cycle6/Day1 (n= 15) | 1670.40 (1614.07)

7. Secondary Outcome: Plasma Trough Concentrations (Ctrough) of Trastuzumab
Description: Ctrough = the concentration prior to study medication administration.
Time Frame: Weekly trastuzumab: Pre-dose (0 H) on Day 1 and 15 of Cycle 1, 2, 4 and 6; 3-weekly trastuzumab: Pre-dose (0 H) on Day 1 of Cycle 1, 2, 4 and 6
Population: Data was not summarized since majority of observed Ctrough values were below lower limit of quantification.
Arm/Group | Sunitinib + Docetaxel + Trastuzumab
Number analyzed (Participants) | 0

8. Other Pre Specified Outcome: Maximum Observed Plasma Concentration (Cmax) of Paclitaxel
Time Frame: End of infusion (1 H) on Day 1 of Cycle 1, 2, 4 and 6
Population: Data not analyzed since paclitaxel was not administered in the study.
Arm/Group | Sunitinib + Docetaxel + Trastuzumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Sunitinib + Docetaxel + Trastuzumab
Serious Adverse Events (participants affected / at risk) | 11/25
Other Adverse Events (participants affected / at risk) | 23/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib + Docetaxel + Trastuzumab (N=25)
Febrile neutropenia (Blood and lymphatic system disorders) | 4
Neutropenia (Blood and lymphatic system disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Multi-organ failure (General disorders) | 1
Erysipelas (Infections and infestations) | 1
Pseudomembranous colitis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1
Syncope (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib + Docetaxel + Trastuzumab (N=25)
Anaemia (Blood and lymphatic system disorders) | 6
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 6
Neutropenia (Blood and lymphatic system disorders) | 14
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Conjunctivitis (Eye disorders) | 5
Lacrimation increased (Eye disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 4
Abdominal pain upper (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 15
Dyspepsia (Gastrointestinal disorders) | 2
Haemorrhoids (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 11
Stomatitis (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 7
Asthenia (General disorders) | 4
Fatigue (General disorders) | 15
Mucosal inflammation (General disorders) | 4
Oedema (General disorders) | 2
Oedema peripheral (General disorders) | 6
Pyrexia (General disorders) | 13
Drug hypersensitivity (Immune system disorders) | 3
Hypersensitivity (Immune system disorders) | 2
Bronchitis (Infections and infestations) | 2
Cystitis (Infections and infestations) | 2
Gastroenteritis viral (Infections and infestations) | 2
Pharyngitis (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 2
Weight decreased (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 8
Dizziness (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 4
Headache (Nervous system disorders) | 4
Paraesthesia (Nervous system disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5
Acne (Skin and subcutaneous tissue disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 6
Dermatitis (Skin and subcutaneous tissue disorders) | 2
Hair colour changes (Skin and subcutaneous tissue disorders) | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 6
Rash (Skin and subcutaneous tissue disorders) | 5
Skin discolouration (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 6
Phlebitis (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.